CLINICAL TRIAL: NCT01134211
Title: Clinical Comparison of Two Daily Disposable Lenses Among Daily Disposable Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-337-C-033
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2011-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- nelfilcon A / filcon II 3 (Other): Nelfilcon A contact lenses worn first, with filcon II 3 contact lenses worn second. Both products worn in both eyes on a daily wear, daily disposable basis for one week each.
  Interventions: Device: nelfilcon A; Device: filcon II 3
- filcon II 3 / nelfilcon A (Other): Filcon II 3 contact lenses worn first, with nelfilcon A contact lenses worn second. Both products worn in both eyes on a daily wear, daily disposable basis for one week each.
  Interventions: Device: nelfilcon A; Device: filcon II 3

INTERVENTIONS:
Device: nelfilcon A — Commercially marketed, single-vision, soft contact lens for daily disposable wear
Device: filcon II 3 — Commercially marketed, single-vision, soft contact lens for daily disposable wear

SUMMARY:
The primary objective of this trial is to evaluate the subjective performance of two different daily disposable contact lenses in a population of daily disposable lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing any spherical daily disposable lens in daily wear, daily disposable modality for at least 3 months prior to enrollment with the exception of the 2 study products
* Currently Wearing lenses at least 8 hrs/day and 5 days/week.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks immediately prior to enrollment for this trial.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in any clinical trial.
* Evidence of systemic or ocular abnormality, infection, or disease which is likely to affect successful wear of contact lenses or use of their accessory solutions as determined by the investigator.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* Prior history of corneal or refractive surgery.
* Requires monovision correction.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
subjective ratings and preferences | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- W.Hartwig - Qualität in jeder Hinsicht, Heikendorf, Germany

REFERENCES:
- [Result] OVS, Marx et al. Subjective Performance of hydrogel and silicone hydrogel daily disposable contact lenses). AAO poster presentation 2014.